CLINICAL TRIAL: NCT00003858
Title: A Phase II Trial of Adjuvant Mitoxantrone (NSC #301739) for High Risk Patients Following Radical Prostatectomy
Brief Title: Mitoxantrone Following Surgery in Treating Patients With Prostate Cancer at High Risk for Recurrence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was not activated.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-99801; CLB-99801; CDR0000067021 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-09-14 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mitoxantrone

ARMS (1):
- Mitoxantrone (Experimental): Patients receive mitoxantrone IV over 10-30 minutes every 21 days. Treatment continues for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for the first 3 years, and then every 6 months for the next 3 years or until disease progression.
  Interventions: Drug: mitoxantrone hydrochloride

INTERVENTIONS:
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy after surgery may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of mitoxantrone given after surgery in treating patients who have prostate cancer that is at high risk for recurrence.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the feasibility of enrolling patients with adenocarcinoma of the prostate at high risk for recurrence following radical prostatectomy in an adjuvant mitoxantrone trial. II. Determine if this adjuvant therapy results in a delay in time to failure or a decrease in the number of treatment failures compared to historical controls in this patient population.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Adenocarcinoma of the prostate treated by radical prostatectomy within the past 3 months Considered to be at high risk for recurrence as defined by at least 1 of the following characteristics on the radical prostatectomy specimen: Positive seminal vesicles Gleason 6 and preoperative PSA greater than 18 ng/mL Gleason 7 and preoperative PSA greater than 14 ng/mL Gleason 8, 9, or 10 and any preoperative PSA Undetectable PSA (i.e., less than 0.1 ng/mL) within 3 months following radical prostatectomy and at time of enrollment Negative lymph nodes at time of radical prostatectomy if lymphadenectomy performed Extracapsular penetration and/or positive surgical margins allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-1 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Not specified Cardiovascular: No New York Heart Association class III or IV cardiac disease or angina pectoris No myocardial infarction within the past 6 months

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent filgrastim or sargramostim except for febrile neutropenia Chemotherapy: No other concurrent chemotherapy Endocrine therapy: No prior neoadjuvant or adjuvant hormonal therapy for prostate cancer No concurrent hormonal therapy except for non-disease related conditions (e.g., insulin for diabetes) No concurrent systemic corticosteriods unless for adrenal insufficiency No concurrent prednisone, dexamethasone, or other steroidal antiemetics At least 6 months since prior finasteride No concurrent finasteride No concurrent antiandrogens (e.g., flutamide, bicalutamide, nilutamide) or gonadotropin releasing hormone agonists (e.g., leuprolide, goserelin) Radiotherapy: No prior adjuvant radiotherapy for prostate cancer No prior pelvic radiotherapy for prostate cancer Surgery: See Disease Characteristics Other: At least 6 months since prior saw palmetto No concurrent compounds with 5 alpha-reductase inhibitor activity (e.g., saw palmetto)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Decrease in time to failure | Up to 3 years

SECONDARY OUTCOMES:
Decrease in the number of treatment failures | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Presti, MD, Study Chair — Stanford University

REFERENCES:
- [Result] Levine EG, Halabi S, Roberts JD, Kaplan EB, Rago R, Atkins JN, Vogelzang NJ. Higher doses of mitoxantrone among men with hormone-refractory prostate carcinoma: a Cancer and Leukemia Group B study. Cancer. 2002 Feb 1;94(3):665-72. doi: 10.1002/cncr.10217. PMID 11857298